CLINICAL TRIAL: NCT01162356
Title: A Prospective Analysis of Nerve Fiber Layer and Macular Changes After Pars Plana Vitrectomy
Brief Title: Prospective Retinal and Optic Nerve Vitrectomy Evaluation (PROVE) Study
Acronym: PROVE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Associate Professor of Ophthalmology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 100073
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma; Macular Pucker; Macula Hole; Vitreomacular Traction; Vitreous Opacities or Hemorrhage
Keywords: Vitrectomy; Glaucoma; Macula; Optic nerve; Ocular Coherence Tomography
MeSH Terms: conditions — Glaucoma; Epiretinal Membrane; Retinal Perforations; vitreous floaters; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Since the introduction of vitrectomy in 1971, this procedure has become the third most frequently performed ophthalmic surgery. Approximately 225,000 vitrectomies are performed annually in the United States and indications continue to expand. Known long-term complications of vitrectomy are relatively few and include retinal detachment and cataract formation. Although much has been written in the literature concerning acute rises in intraocular pressure (IOP) in the immediate postoperative period, there is surprisingly little information on long term IOP outcomes after vitrectomy. A recent report by Chang given at the LXII (62) Edward Jackson Memorial Lecture hypothesized a causal relationship between vitrectomy and open-angle glaucoma (OAG) via oxidative stress exacerbated by removal of the crystalline lens. A second report by Luk and colleagues reported similar conclusions in a modified cohort. Both studies, were retrospective in nature and did not perform baseline evaluations to exclude pre-existing glaucoma. Furthermore neither study accounted for natural history. Finally, our analysis has not reproduced similar results.

The primary purpose of this study is to analyze the full spectrum of optic nerve and macular changes between vitrectomized study eyes and their non-vitrectomized fellow eyes to control for natural history. Baseline evaluations will include examination by fellowship trained retina and glaucoma specialists, fundus photography, autofluorescence, optical coherence tomography (macula and optic nerve) and automated visual field testing. At 3 month then annually for 5 years after vitrectomy surgery, the cohort will undergo similar evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent and comply for the duration of the study and imaging studies
* Media clarity sufficient for imaging studies
* No previous treatment or surgery that might confound study results in the study or fellow eye
* Pars plana vitrectomy (PPV) indicated for epiretinal membrane (ERM), macular hole (MH), vitreo-macular traction (VMT), and vitreous hemorrhage (VH)

Exclusion Criteria:

* Unable to consent and/or comply for the duration of the study and imaging studies
* History of the following conditions: Glaucoma or associated conditions, visual field defects, uveitis, age-related macular degeneration (ARMD), prior PPV for retinal detachment, retained lens or dislocated intraocular lens
* Contralateral eye status post PPV or with advanced eye disease serious enough to warrant future PPV - Contralateral eye with condition that may result in choroidal neovascular membrane

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to ophthalmology practice requiring pars plana vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Nerve fiber layer and macular changes after vitrectomy | 3 month and annually for 5 years after surgery
  To determine the incidence of nerve fiber layer (NFL) and macular changes after pars plana vitrectomy, characterize their extent and quality, and determine pre-disposing risk factors.

SECONDARY OUTCOMES:
Visual field defects | 3 month and annually for 5 years after surgery
  To characterize long-term functional consequences of NFL or macular changes with regards to peripheral and central visual field defects after PPV.
Open-angle glaucoma | 3 month and annually for 5 years after surgery
  To determine the incidence of elevated intraocular pressure and open-angle glaucoma following vitrectomy. Enrolled patients will be screened at baseline to exclude pre-existing glaucoma and post-operative glaucoma screenings will be performed by fellowship trained glaucoma specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt Eye Institute; Maziar Lalezary, MD, Study Director — Vanderbilt Eye Institute; Rahul K Reddy, MD, Study Director — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

REFERENCES:
- [Background] Machemer R, Buettner H, Norton EW, Parel JM. Vitrectomy: a pars plana approach. Trans Am Acad Ophthalmol Otolaryngol. 1971 Jul-Aug;75(4):813-20. No abstract available. PMID 5566980
- [Background] Chang S. LXII Edward Jackson lecture: open angle glaucoma after vitrectomy. Am J Ophthalmol. 2006 Jun;141(6):1033-1043. doi: 10.1016/j.ajo.2006.02.014. PMID 16765671
- [Background] Luk FO, Kwok AK, Lai TY, Lam DS. Presence of crystalline lens as a protective factor for the late development of open angle glaucoma after vitrectomy. Retina. 2009 Feb;29(2):218-24. doi: 10.1097/IAE.0b013e31818ba9ca. PMID 18936722